CLINICAL TRIAL: NCT04972838
Title: Autism Intervention Research Network on Behavioral Health: Remaking Recess
Brief Title: AIR-B4: Remaking Recess (RR)
Acronym: RR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Collaborators: University of California, Davis (Other); University of Kansas (Other); University of Washington (Other); University of Pennsylvania (Other); University of Rochester (Other); Drexel University (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor of Human Development and Psychology, Health Resources and Services Administration (HRSA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-001993
Record Dates: First submitted 2021-07-06; First posted 2021-07-22 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder; Neurodevelopmental Disorders
Keywords: autism; playground; recess; inclusive school culture
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UNITED (Experimental): UNITED is premised on the idea that successful implementation in organizations like schools and early intervention systems requires a team-based approach, in which the team is thoughtfully assembled, develops a plan for implementation, assigns roles and responsibilities, and carefully tracks and supports implementation and sustainment in all its stages within a few meetings and ongoing coaching from the research staff.
  Interventions: Behavioral: Remaking Recess (RR)
- Implementation as Usual (IAU) (Active Comparator): The organizations will implement RR as usual. The research team will be available to provide support on the RR intervention as needed.
  Interventions: Behavioral: Remaking Recess (RR)

INTERVENTIONS:
Behavioral: Remaking Recess (RR) — Remaking Recess is a flexible, school-based social engagement intervention for students with autism and their peers. The research team will work with school personnel to deliver RR during recess. RR is tailored based on the needs of schools, students, and staff.

SUMMARY:
The AIRB research team will compare the use and effectiveness of each intervention (Mind the Gap, Remaking Recess and Self Determination Learning Model of Instruction) with and without the addition of our implementation strategy, UNITED. In all groups, the research team will train community practitioners using remote delivery of professional development modules specific to the intervention, and active coaching for up to 12 sessions as dictated by the intervention procedures.

The research team will pair UNITED with three interventions that cover the ages of early childhood, childhood, and adolescence. These include Mind the Gap (MTG), a family navigation intervention for children newly diagnosed under age 8, Remaking Recess (RR), a school-based social/peer engagement intervention for children ages 5-12, and Self-Determination Learning Model of Instruction (SDMLI), a self- advocacy intervention for adolescents (13-22 years; 22 is the upper age limit of high school for individuals with disabilities).

For Remaking Recess, school personnel will be working with children with ASD using the Remaking Recess Intervention (play-based intervention done during recess). School personnel will be trained to implement the intervention. The total time commitment for the school personnel is about 30 hours. The total time commitment for the parents with ASD who will sign consents and fill out a demographic survey is about 15 minutes. The total time commitment for children with ASD or other neurodevelopmental disorders (NDD) is about 5 hours during their regularly scheduled recess period throughout the school year.

DETAILED DESCRIPTION:
Remaking Recess (RR) will include 112 elementary school personnel (e.g., playground staff, classroom aides, teachers); and 152 children with ASD/NDD ages 5-12 (2-5 per school).

RR targets school staff on the recess yard who supervise all students, including those with ASD/NDD. Training in RR will be remote, with all schools receiving a 60-90 minute didactic training during district professional development days which has been successful in previous studies. Active coaching (via remote methods, most likely zoom) will occur weekly with staff at school for 10-12 sessions during RR implementation with enrolled students. In prior studies, various school personnel (e.g., teachers, counselors, bus attendants, noontime aides, classroom assistants, and one-to-one paraprofessionals) have served as intervention agents.

There will be 3 assessment time points. At entry, the teachers/school staff will fill out Demographic, Implementation Climate Scale, Teacher perceptions, Clinical Global Impression (CGI-I), Social Network survey, and fidelity forms. The Staff Diary will be completed on an ongoing basis coinciding with coaching sessions. At the midpoint of the study (midpoint of school year) and at exit (end of the school year), they will fill out Implementation Climate Scale, Teacher perceptions, Clinical Global Impression (CGI-S, CGI-I), Social Network survey, and fidelity forms. The Social Network survey will be completed once in the following school year.

All participants in RR will be randomized to receive UNITED, exploratory implementation strategy, or implementation as usual (IAU). UNITED is premised on the idea that successful implementation in organizations like schools and early intervention systems requires a team-based approach, in which the team is thoughtfully assembled, develops a plan for implementation, assigns roles and responsibilities, and carefully tracks and supports implementation and sustainment in all its stages. To address these requirements, the research team combined two well-tested strategies. The first is social network analysis (SNA) through which we will systematically identify members of the team who will implement each intervention. The second is TeamSTEPPS (Team Strategies and Tools to Enhance Performance and Patient Safety), an evidence-based set of teamwork tools that optimizes target population outcomes by improving communication and teamwork skills. The research staff will approach the school leaders (2 at maximum) and explain Remaking Recess. After the school leaders agree to participate in the study, they will complete a site agreement to participate and then fill out the Social Network Assessment (SNA) to provide names, roles, and emails of staff at the agency that have significant roles in the school that relate to the Remaking Recess intervention. The research staff will then email these school personnel the SNA as well. After receiving the completed SNA assessments, the research team will randomize each organization to UNITED vs Implementation as Usual (IAU). The research team will use the data from these assessments to assess both arms of the study. Additionally, for those randomized to UNITED, Dr. Elizabeth McGhee Hassrick at Drexel University and her team, will provide the research sites the top 2-5 school personnel identified by the SNA as key for intervention implementation support. This team will be invited to participate in the UNITED implementation team. If they agree, they will complete a School Personnel Consent (UNITED/IAU) before beginning any UNITED training. For both UNITED and IAU schools, the school personnel that will be implementing Remaking Recess will fill out the Remaking Recess School Personnel Consent (Implementor) before beginning any study procedures.

ELIGIBILITY:
Inclusion Criteria:

* 112 elementary school personnel ( e.g. playground staff, classroom aides, teachers)
* 152 children with ASD or NDD ages 5 to 12 and family is under-resourced.
* Expert medical diagnosis or educational classification of ASD
* Spend majority of the day (51%) in a general education classroom

Under-resourced, defined by:

* Attending a Title I school (a school that receives federal funding to improve the performance of economically disadvantaged students)or rural school
* Family income is under 250% of the federal guidelines for poverty rate (i.e., meets federal requirements to qualify for free or reduced lunch)
* Parent/Caregiver willing to participate

Exclusion Criteria:

* Personnel at school not working with children with ASD or NDD Children: Under the age of 5 or over 12, does not spend majority of the day (51%) in general education classroom, does not have ASD or NDD and family is not under-resourced.

No official ASD/NDD diagnosis. Parent/Caregiver not willing to participate.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 264 (Estimated)
Dates: Start 2021-07-11 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Stages of Implementation Completion (SIC) | through study completion, an average of 18 months
  ool developed by the Oregon Social Learning Center, is an 8 stage tool of implementation process and milestones, with stages spanning three implementation phases (pre-implementation, implementation, and sustainability.

SECONDARY OUTCOMES:
School Implementation Climate Scale | baseline,12 weeks, and 24 weeks
  This scale was adapted to be used by the research team to gather information from the schools/agencies in the study about the use of evidence-based practices in their organizations. It is scaled from 0(not at all) to 4 (very great extent). Higher scores mean better outcomes.
Social Network Survey- participants of survey will name key personnel that can be participants of the UNITED team for this intervention | baseline, 12 months, and 18 months
  Survey created by the research team to gather information about the key people in each organization that can better support the Remaking Recess intervention.
Teacher Perceptions Scale | baseline, 12 weeks, and 24 weeks
  Survey adapted by the research team to better understand the target student's behavior in the classroom and with his/her peers. It is rated using 1 as never, 2 as sometimes, and 3 as very often, with "3" as showing better outcome.
Clinical Global Rating (CGI) | baseline, 12 weeks, and 24 weeks
  Survey created by the research team to show how the child is doing in terms of his/her social functioning. It is rated from "1" to "7", with "1" being "typical" and showing better outcomes and "7" as "extreme" and showing lowest outcome.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Rochester, Rochester, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Locke J, Hassrick EM, Stahmer AC, Iadarola S, Boyd B, Mandell DS, Shih W, Hund L, Kasari C; AIR-B Network. Using Novel Implementation Tools for Evidence-based Intervention Delivery (UNITED) across public service systems for three evidence-based autism interventions in under-resourced communities: study protocol. BMC Psychiatry. 2022 Jul 16;22(1):478. doi: 10.1186/s12888-022-04105-9. PMID 35842614